CLINICAL TRIAL: NCT06233370
Title: Acute Effects of Walking Exercise on Brain Functioning in Multiple Sclerosis
Acronym: PRIMERS
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Brian Sandroff, Senior Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: R-1234-23
Record Dates: First submitted 2023-12-18; First posted 2024-01-31 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
Keywords: exercise; MRI; walking
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will complete two single bouts of walking exercise. One bout of walking exercise involves walking at a moderate intensity over ground, and the other bout of walking exercise involves walking at a moderate intensity on a treadmill. The order of walking exercise bouts will be randomly determined and counterbalanced across participants. Before and after each bout of walking exercise, participants will complete an MRI scan to measure brain connectivity and brain blood flow.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Over ground walking exercise (Experimental): Participants will walk around a square hallway at a step rate of ~100 steps per minute for 20 minutes while wearing a Fitbit around the waist for measuring steps.
  Interventions: Behavioral: Moderate intensity walking exercise
- Treadmill walking exercise (Experimental): Participants will walk on a motor-driven treadmill at a step rate of ~100 steps per minute for 20 minutes while wearing a Fitbit around the waist for measuring steps.
  Interventions: Behavioral: Moderate intensity walking exercise

INTERVENTIONS:
Behavioral: Moderate intensity walking exercise — For each intervention arm, participants will be walking at a moderate intensity, determined based on a step rate of approximately 100 steps per minute (measured by a Fitbit)

SUMMARY:
The project will involve a within-subjects, repeated-measures research design. Participants will initially be screened for relevant inclusion/exclusion criteria for maximizing safety of participating in an exercise study. If a participant meets those inclusion/exclusion criteria, they will visit Kessler Foundation three times. The first visit will involve a baseline session where participants will complete several cognitive tests. This will be followed by a training session, where participants will be provided with a FitBit, and will be trained by research staff to walk at a rate of 100 steps per minute. Once participants demonstrate proficiency at walking at this rate using the FitBit, participants will complete several questionnaires, followed by a maximal, graded exercise test to determine cardiorespiratory fitness. One week later, participants will return to Kessler Foundation to complete 1 of 2 experimental sessions that will be delivered in a random order that further will be counterbalanced across participants (to minimize the potential effects of session order on brain function and blood flow, respectively). Both experimental sessions will follow the same structure. First, participants will undertake a 30-minute MRI scan at Kessler Foundation to measure brain function and brain blood flow. Immediately following the MRI scan, participants will engage in either 20 minutes of treadmill walking exercise or 20 minutes of overground walking exercise at a rate of 100 steps per minute. Immediately following the 20-minute exercise bouts, participants will undertake another MRI scan for measuring brain function and brain blood flow. Participants will return to Kessler Foundation a third time to complete the opposite experimental session that was not completed during the second visit (i.e., overground walking exercise if treadmill walking exercise was completed during the second visit). In total, each participant will undergo four MRI scans over the course of the study (i.e., pre-treadmill, post-treadmill, pre-overground, post-overground). .

ELIGIBILITY:
Inclusion Criteria:

* Clinically-definite MS diagnosis
* Relapse-free for at least 30 days
* Low risk for contraindications for exercise testing
* Low risk for contraindications for MRI
* Historically physically inactive prior to MS diagnosis
* Historically highly physically active prior to MS diagnosis

Exclusion Criteria:

* Diagnosis of uncontrolled major depressive disorder, schizophrenia, bipolar disorder I or II, or substance use disorders
* Taking medications that can affect cognition (e.g., antipsychotics, benzodiazepines)
* Historically moderately physically active prior to MS diagnosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain Function | Weeks 2 and 3
  MRI-measured resting-state functional connectivity of the thalamus with other areas of the brain
Brain Blood Flow | Weeks 2 and 3
  MRI-measured cerebral blood flow perfusion in the left and right hemispheres

OTHER OUTCOMES:
Aerobic fitness | Week 1
  Cardiorespiratory fitness (i.e., peak oxygen consumption (VO2peak)) based on a maximal graded exercise test on a motor-driven treadmill
Average steps per day | Week 1
  Free-living physical activity based on average steps per day measured by an ActiGraph accelerometer for a 7-day period
Cognitive processing speed | Week 1
  Performance on the Symbol Digit Modalities Test (raw score). Higher scores are indicative of faster cognitive processing speed
Aerobic fitness | Week 1
  Cardiorespiratory fitness (i.e., time to exhaustion) based on a maximal graded exercise test on a motor-driven treadmill
Verbal learning and memory | Week 1
  Performance on the California Verbal Learning Test II (raw score). Higher scores are indicative of better learning and memory
Visuospatial learning and memory | Week 1
  Performance on the Brief Visuospatial Memory Test-Revised (raw score). Higher scores are indicative of better visuospatial learning and memory
Time spent in moderate-to-vigorous physical activity | Week 1
  Free-living physical activity based on time spent in moderate-to-vigorous activity measured by an ActiGraph accelerometer for a 7-day period

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will share de-identified IPD upon request for inclusion in potential meta-analyses